CLINICAL TRIAL: NCT03948529
Title: RevErsing Poor GrAft Function With eLtrombopag After allogeneIc Hematopoietic Cell trAnsplantation: a Prospective, Phase II Study by the SFGM-TC
Brief Title: RevErsing Poor GrAft Function With eLtrombopag After allogeneIc Hematopoietic Cell trAnsplantation
Acronym: REGALIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: inclusions difficulties.
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017_52; 2018-001157-27 (EudraCT Number)
Record Dates: First submitted 2019-02-28; First posted 2019-05-14 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Leukemia; Graft Failure
Keywords: Poor Graft Function (PGF),; Allogeneic hematopoietic cell transplantation (Allo-HCT); Eltrombopag.
MeSH Terms: conditions — Leukemia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eltrombopag (Experimental): Eligible patients will receive the investigational drug eltrombopag
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — eltrombopag at the starting dose of 50mg/day. After 2 weeks of eltrombopag initiation and in the absence of platelet response, eltrombopag will be increased every two weeks (50mg increase) up to a maximum dose of 150mg/day (2 maximum escalation from D1, with maximum dose escalation phase of 4 weeks).

SUMMARY:
Poor graft function (PGF) after allogeneic hematopoietic cell transplantation (allo-HCT) is a misunderstood complication associated with poor outcome and limited therapeutic options. Despite the lack of standardized diagnostic criteria, PGF is commonly defined as follows: one or several significant cytopenias after allo-HCT persisting or developing after allo-HCT despite full donor chimerism and in the absence of relapse or other causes. Not only PGF can alter patients' quality of life by leading to recurrent transfusions, bleeding events and infections, but it is also associated with poor survival after allo-HCT.

Although PGF is relatively frequent, there is no well-codified behavior in the literature or in the recommendations issued by the various learned societies of transplantation.

The aim objective of the investigator's study is to demonstrate that eltrombopag improve PGF after allo-HCT

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of poor graft function defined as:

  * Patient ≥ day+60 after allo-HCT,
  * Persisting thrombocytopenia on two different samples over at least two weeks (platelet < 30G/L with transfusion requirement) +/- neutropenia (ANC <1G/L) +/- anemia (Hb <8g/dL or transfusion requirement),
  * Full donor chimerism on whole blood (≥ 95%),
  * Biopsy proven hypocellular marrow without evidence of myelodysplasia
  * No evidence for relapse,
  * No evidence for active acute or chronic graft versus host disease,
  * Absence of active viral infection (EBV, CMV, ADENOVIRUS, PARVOVIRUS B19),
  * Absence of B9/B12 deficiency,
  * Absence of hypothyroidism,
  * Absence of hypogonadism,
  * Absence of dialysis,
  * Absence of thrombotic microangiopathy,
  * Absence of macrophage activation syndrome,
  * No other known causes of poor graft function.
* Written informed consent must be obtained before any study-trial specific procedure are performed,
* Affiliation to a social security system.

Exclusion Criteria:

* Criteria for poor graft function not fulfilled (see above),
* Patients aged less than 6 years old (or unable to swallow),
* Hepatic impairment (Child-Pugh ≥ 5),
* Patients with bone morrow fibrosis,
* Patients with a cytogenetic abnormality of chromosome 7
* Hypersensitivity to eltrombopag or to any of the excipients,
* Patients with any contra-indication to eltrombopag, filgrastim,
* Unable to understand the investigational nature of the study or give informed consent,
* History of congestive heart failure, arrhythmia requiring chronic treatment, arterial or venous,
* Thrombosis (not excluding line thrombosis) within the last 1 year, or myocardial infarction within 3 months before enrollment,
* ECOG Performance Status of 3 or greater,
* Pregnant and/or lactating women,
* Freedom privacy.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Platelet response | at 12 weeks
  Platelet response defined as a platelet count ≥ 30G/L at 12 weeks measured on at least two serial measurements performed 1 week apart and sustained for 1 month or more without support of platelet transfusions.

SECONDARY OUTCOMES:
Time to erythroid response | at 12 and 24 weeks
  Time to erythroid response defined as an increase of at least 1.5g/dL without transfusion, that is sustained for at least 2 weeks and transfusion requirements at 12 and 24 weeks for BRC as compared with transfusion requirements during the eight weeks preceding study entry
Time to neutrophil response | at least 7 days
  Time to neutrophil response defined as an increase of ANC above 1G/L, which is sustained for at least 7 days,
Percentage of patients presenting best bone marrow response at 12 and 24 weeks of treatment assessed by bone marrow aspirate and bone marrow biopsy with fibrosis staining. | at 12 and 24 weeks
Transfusion requirements | at 12 and 24 weeks
  Transfusion requirements for BRC and platelets as compared with transfusions requirements during the eight weeks preceding study entry
Proportion of patients presenting grade 3 or 4 adverse events from the first to the last administration of eltombopag. | from 1st administration of eltrombopag to 1 month after the last administration of eltrombopag,
  All adverse events will be reported on the adverse events reporting form of the case report file. Each adverse event will be recorded individually.
  The severity of the adverse event will be determined as follows :
  * Severe (grade 3): significant interference with the patient's daily activity and unacceptable,
  * Life-threatening (grade 4).
Quality of life evaluation using the European Organisation for Research Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30 questionnaire). | at 12 and 24 weeks
  The QLQ-C30 consists of thirty items:
  * 05 functional scales to explore the physical (1 to 5), executive (6 to 7), social (26 and 27), cognitive (20 and 25), and emotional (21 to 24) dimensions of the quality of life.
  * 09 symptomatic scales to explore fatigue (10, 12 and 18), nausea symptoms (14 and 15), pain (9 and 19), dyspnea (8), insomnia (11), anorexia (13), diarrhea (17), constipation (16) and financial difficulties (28).
  * 01 scale measuring the overall quality of life of each patient (29 and 30). The results of these different scales allow the calculation of a score that varies from 0 (worst) to 100 (better). A high overall health score reflects good health and a good quality of life. A high score for a symptom scale reflects a high level of symptoms. An average difference of 5 to 10 scores between two visits indicates a minor change, from 10 to 20 a moderate change and a difference of more than 20 points a significant change.
Immune function (T/B/NK cells counts) | at 12 and 24 weeks
Overall survival, relapse-free survival and non-relapse mortality | at 24 weeks of treatment
  No relapse disease will be investigated using the Fine-Gray Test. No relapse mortality represent all death without relapse of the underlind disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Yakoub-Agha, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France